CLINICAL TRIAL: NCT00743795
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Trial Comparing 24 or 48 Weeks of GS 9190, in Combination With Peginterferon Alfa 2a and Ribavirin, to 48 Weeks of Peginterferon Alfa 2a and Ribavirin for the Treatment of Genotype-1 Chronic Hepatitis C Virus (HCV) Infection (GS-US-196-0103)
Brief Title: Safety, Tolerability, and Antiviral Activity of 24 or 48 Weeks of GS-9190 in Combination With Peginterferon Alfa 2a and Ribavirin for the Treatment of Genotype-1 Chronic HCV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-196-0103
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-10

CONDITIONS: HCV Infection
Keywords: Hepatitis C; HCV; Rapid Virologic Response; Sustained Virologic Response; HCV RNA; Polymerase inhibitor; GS-9190
MeSH Terms: conditions — Hepatitis C | interventions — tegobuvir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): Peginterferon and ribavirin + placebo BID for 48 weeks + 24 weeks treatment-free follow-up (n = 50)
  Interventions: Drug: placebo; Drug: Peginterferon Alfa 2a; Drug: Ribavirin
- 2 (Experimental): Peginterferon and ribavirin + GS 9190 40 mg BID for 48 weeks + 24 weeks treatment-free follow-up (n = 100)
  Interventions: Drug: GS-9190; Drug: Peginterferon Alfa 2a; Drug: Ribavirin
- 3 (Experimental): Peginterferon and ribavirin + GS 9190 40 mg BID for 48 weeks + 24 weeks treatment-free follow-up. However, subjects who achieve RVR (HCV RNA undetectable at Week 4) and maintain that response through Week 24 will stop all study drugs at Week 24 and be followed for an additional 48 weeks (n = 50).
  Interventions: Drug: GS-9190; Drug: Peginterferon Alfa 2a; Drug: Ribavirin

INTERVENTIONS:
Drug: placebo — oral BID
  Arms: 1
Drug: GS-9190 — 40 mg oral BID
  Arms: 2; 3
Drug: Peginterferon Alfa 2a — All subjects received a fixed dose of 180 μg PEG via subcutaneous injection on a weekly basis.
  Other Names: PEG
Drug: Ribavirin — Ribavirin supplied as 200 mg Copegus® tablets (1000 mg for subjects weighing < 75 kg and 1200 mg for subjects weighing ≥ 75 kg) were given in a divided daily dose.
  Other Names: RBV

SUMMARY:
The purpose of this study is to compare the safety, tolerability and effectiveness of the experimental drug GS-9190 when administered for 24 or 48 weeks with peginterferon alfa 2a and ribavirin for the treatment of genotype-1 chronic hepatitis C infection.

DETAILED DESCRIPTION:
The safety, tolerability and antiviral efficacy GS-9190, administered orally twice daily at 40 mg, will be compared to placebo when used in combination with peginterferon alfa 2a (PEG) and ribavirin (RIBA) in treatment-naïve subjects chronically infected with HCV genotype 1 infection. Two-hundred forty-eight (248) subjects will be randomized (ratio: 1:2:1) to one of three treatment arms:

Arm 1: PEG/RIBA + placebo BID for 48 weeks + 24 weeks treatment-free follow-up (n = 62)

Arm 2: PEG/RIBA + GS 9190 40 mg BID for 48 weeks + 24 weeks treatment-free follow-up (n = 124)

Arm 3: PEG/RIBA + GS 9190 40 mg BID for 48 weeks + 24 weeks treatment-free follow-up. However, subjects who achieve RVR (HCV RNA undetectable at Week 4) and maintain that response through Week 24 will stop all study drugs at Week 24 and be followed for an additional 48 weeks (n = 62).

Randomization will be stratified by plasma HCV RNA level (< or ≥ 400,000 IU/mL) at screening and race (of African descent or other).

In order to ensure adequate representation of subjects with genotypes 1a and 1b in this trial, enrollment for either genotype will be capped at 120 subjects. Once 120 subjects of either genotype (e.g., genotype 1a) have been randomized, subsequent enrollment will only be allowed for subjects with the other genotype (e.g., genotype 1b).

The duration of double-blind treatment is 48 weeks plus 24 weeks of treatment-free follow-up; however subjects in Arm 3 will stop all medication at Week 24 if they have achieved an RVR (defined by undetectable HCV RNA following 4 weeks on therapy) and have maintained that response thereafter. Subjects will only learn that they have been randomized to Arm 3 if, at Week 24, having achieved criteria for stopping therapy, they are instructed to stop. All other subjects will remain blinded to their treatment status throughout the course of the study.

The standard of care treatment stopping criterion used in clinical practice when treating HCV with PEG/RIBA, failure to achieve EVR, will be utilized in this trial. Additionally, subjects with detectable plasma HCV RNA at Week 24 will discontinue all study medications no later than the Week 28 visit and will be followed off-treatment for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18 - 70 years of age)
* Chronic HCV infection for at least 6 months prior to Baseline (Day 1) (anti-HCV antibody positive; positive for plasma HCV RNA; medical history consistent with chronicity accepted by the investigator)
* Liver biopsy results within the past 2 years prior to Baseline (Day 1) indicating the absence of cirrhosis
* HCV treatment-naive, defined as no prior exposure to PEG, RIBA, or experimental HCV therapy
* Mono-infection with HCV genotype 1a or 1b
* Detectable plasma HCV RNA at Screening
* BMI between 19 and 36 kg/m2
* Willing and able to provide written informed consent and to comply with all study requirements
* Of generally good health as determined by the Investigator
* Subject agrees to use adequate skin protection (e.g., sunblocking agent) when exposed to the sun.
* Women of childbearing potential (i.e., a non-menopausal female or a female with menopausal < 2 years, who has not had a hysterectomy, bilateral oophorectomy or medically documented ovarian failure) must have negative serum β-human chorionic gonadotropin (hCG) at screening and negative urine pregnancy test prior to the first study drug administration.
* All subjects (male and female) must agree to utilize highly effective contraception methods (two separate forms of contraception, one of which must be an effective barrier method, or be non-heterosexually active, practice sexual abstinence or have a vasectomized partner) from screening throughout the duration of study treatment and for 24 weeks after the last dose of RIBA.
* Female subjects who utilize hormonal contraceptive as one of their birth control methods must have used the same method for at least three months prior to study dosing.
* Female subjects who are postmenopausal for less than two years are required to have FSH > 40 mIU/mL. If the FSH is ≤ 40 mIU/mL, the subject must agree to use highly effective method of birth control (as described above) to participate in the study.
* Male subjects who are sexually active must be willing to use effective barrier contraception (e.g., condom with spermicide) during heterosexual intercourse from screening through completion of the study and continue for 24 weeks after the last dose of RIBA

Exclusion Criteria:

* Pregnant or breast feeding women or women who may wish to become pregnant during the course of the study
* Males who have partners planning to become pregnant
* Males and females of reproductive potential who are unwilling to use two forms of effective birth control through Study Week 72. One method should include a condom with spermicide for males
* Infection with non-genotype 1 HCV
* Poorly controlled diabetes mellitus (hemoglobin A1c > 7) unless treatment intervention has been reviewed with the Medical Monitor and improved glucose control is anticipated
* History of sarcoidosis
* History of hemoglobinopathy (e.g., thalassemia)
* History of known retinal disease
* History of invasive malignancy diagnosed or treated within 5 years (recent localized treatment of squamous or non-invasive basal cell skin cancers is permitted; cervical carcinoma in situ is allowed if appropriately treated prior to screen)
* Evidence of hepatocellular carcinoma
* Chronic liver disease of a non-HCV etiology
* Untreated or significant psychiatric illnesses including severe depression, schizophrenia, psychosis, or a history of a suicide attempt
* Co-infection with HIV, HBV, or multiple HCV genotypes
* Chronic use of systemic immunosuppressive agents
* Presence of autoimmune disorders. Subjects with treated hypothyroidism with normal TSH may be enrolled.
* Severe chronic obstructive pulmonary disease
* History of clinically significant cardiac disease, including a family history of Long QT Syndrome, and/or evidence of the following ECG abnormalities at screening: QTcF (QT corrected using Fridericia's formula) of > 450 msec; complete or incomplete left or right bundle branch block; intraventricular conduction delay with QRS duration of > 120 msec; bradycardia (< 45 beats per minute); pathologic Q-waves (Q wave of > 40 msec or depth of > 0.4 to 0.5 V); arrhythmia (an isolated premature ventricular contraction on screening/Day 1 is not exclusionary) ; ventricular pre excitation; second or third degree heart block
* Positive urine screen for amphetamines or cocaine
* Known, current heroin, morphine, or methadone use
* Ongoing alcohol abuse in the judgment of the investigator (in no case intake of more than 28 units of alcohol per week [1 unit = ½ pint of beer, 1 glass of wine, 1 shot of spirits])
* Receiving a known potent CYP 3A4 inhibitor within 2 weeks of study drug dosing or are expected to receive such therapy during the course of study drug dosing
* Known hypersensitivity to the study drugs, their metabolites or formulation excipients
* In the judgment of the Investigator, should not participate in the study due to potential clinical or compliance issues

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Undetectable HCV RNA level | At Week 12 for Early Virologic Response (EVR)

SECONDARY OUTCOMES:
Safety and tolerability | Throughout 72 week study period
Undetectable HCV RNA level | Week 4, Week 24 and Week 48
GS-9190 plasma concentrations | Through Week 48
Undetectable HCV RNA | At Week 72 for sustained virologic response (SVR)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Knox, Study Chair — Gilead Sciences
Locations (60):
- United States (40):
  - Anaheim, California
  - Los Angeles, California
  - Newport Beach, California
  - San Clemente, California
  - San Diego, California
  - San Francisco, California
  - Englewood, Colorado
  - Miami, Florida
  - North Miami Beach, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Chicago, Illinois
  - Bowling Green, Kentucky
  - Baton Rouge, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - St Louis, Missouri
  - Cedar Knolls, New Jersey
  - Johnson City, New York
  - New York, New York
  - Plainview, New York
  - Syracuse, New York
  - Asheville, North Carolina
  - Durham, North Carolina
  - High Point, North Carolina
  - Cincinnati, Ohio
  - Tulsa, Oklahoma
  - Philadelphia, Pennsylvania
  - Germantown, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Annandale, Virginia
  - Fairfax, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
- Belgium (4):
  - Brussels
  - Ghent
  - Leuven
  - Liège
- Germany (6):
  - Berlin
  - Cologne
  - Frankfurt
  - Hamburg
  - Hanover
  - München
- Dublin, Ireland
- Poland (6):
  - Bialystok
  - Bydgoszcz
  - Chorzów
  - Czeladź
  - Krakow
  - Warsaw
- Santurce, Puerto Rico
- United Kingdom (2):
  - Birmingham
  - London